CLINICAL TRIAL: NCT04850040
Title: An Efficacy and Safety Study of Camrelizumab in Combination With Apatinib Mesylate and Oxaliplatin for Neoadjuvant Therapy in Patients With Potentially Resectable Hepatocellular Carcinoma.
Brief Title: A Neoadjuvant Hepatocellular Carcinoma Study of Camrelizumab in Combination With Apatinib and Oxaliplatin
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, JIANPING XU, Associate Chief Physician, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC2841
Record Dates: First submitted 2021-04-14; First posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Hepatocellular Carcinoma Resectable
MeSH Terms: interventions — apatinib; camrelizumab; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab+Apatinib Mesylate+Oxaliplatin (Experimental): An study of Camrelizumab in combination with Apatinib Mesylate and Oxaliplatin for neoadjuvant therapy in patients with potentially resectable hepatocellular carcinoma.
  Interventions: Drug: Apatinib Mesylate; Drug: Camrelizumab; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Apatinib Mesylate — 250 mg, oral every other day. Approximately half an hour after a meal (the daily dose should be taken at the same time as possible) with warm boiled water.
Drug: Camrelizumab — 200 mg, 30 minutes intravenous drip (overall dosing time no shorter than 20 minutes and no longer than 60 minutes, including tube flush time) once every 2 weeks, with the first dose administered concurrently with Apatinib Mesylate Tablets.
Drug: Oxaliplatin — 85 mg/m2, once every 2 weeks, to be administered half an hour after Camrelizumab injection.

SUMMARY:
This is a prospective, single-arm, single-center, clinical research.This trial will explore the efficacy and safety of Camrelizumab in combination with Apatinib Mesylate and Oxaliplatin for neoadjuvant therapy in patients with potentially resectable hepatocellular carcinoma.

DETAILED DESCRIPTION:
There is no high-level evidence on the efficacy of systemic therapy in neoadjuvant studies for hepatocellular carcinoma, and guidelines recommend TACE as the treatment of choice. Given that combination therapies such as immunotherapy in combination with targeted therapy and immunotherapy in combination with chemotherapy have achieved good efficacy in systemic therapy for liver cancer, this study is intended to explore the efficacy of TACE.

In this study, we propose to explore the use of kareliozumab in combination with apatinib and oxaliplatin for the treatment of hepatocellular carcinoma.

In this study, we propose to investigate the efficacy and safety of neoadjuvant therapy with kalilizumab in combination with apatinib and oxaliplatin in patients with potentially resectable hepatocellular liver cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-70 years old, both genders.
2. ECOG PS 0-1 points.
3. Hepatocellular liver cancer with a clinical diagnosis consistent with primary hepatocellular liver cancer and a lesion consistent with the Primary Liver Cancer Diagnostic and Treatment Standards (2019) Edition.
4. The hepatobiliary MDT of Cancer Hospital of Chinese Academy of Medical Sciences (MDT) discussed the case as potentially resectable requiring neoadjuvant chemotherapy.
5. Locally advanced, potentially resectable tumors. Ruptured liver tumor or adjacent organ invasion without extrahepatic metastasis (imaging confirmed).

Hepatocellular carcinoma combined with cancerous thrombus in a branch of a grade 1 or 2 vasculature (portal vein, hepatic vein, bile duct) (imaging confirmed).

Lymph node metastasis (image confirmed). Liver tumor ≥ 5 cm; multiple tumors with ≤ 3 tumors, but located in one lobe (imaging [CT, MRI or ultrasound]) Hepatocellular carcinoma tumors located in the middle lobe (segment IV, V, VIII) or caudal lobe of the liver; hepatocellular carcinoma tumors within 1 cm of a branch of a grade 1 or 2 vasculature (portal vein, hepatic vein, bile duct) or involving the above-mentioned vasculature (expected cut edge < 1 cm).

Tumor with satellite foci or subfoci. Tumor without envelope or incomplete tumor with envelope, multi-nodal fusion. 6. NRS ≤3 points. 7. Patients who have not received any previous antineoplastic drug treatment. 8. At least 1 measurable lesion that meets RECIST 1.1 criteria. 9. Liver function Child-Pugh score: grade A-B (≤7). 10. Expected survival > 3 months. 11. Relevant indicators meet the following criteria:

1. blood routine examination HB≥90 g/L； ANC≥1.5×109/L； PLT≥75×109/L；
2. CMP ALB ≥30g/L； ALT and AST< 2.5ULN； TBIL ≤1.5 ULN； Cr ≤1.5ULN 12. Women of childbearing age (18-49 years covered by this protocol) must have a negative pregnancy test (serum or urine) result within 14 days prior to enrollment and voluntarily use an appropriate method of contraception during the observation period and for 8 weeks after the last dose of study drug; for men, they should be surgically sterilized or agree to use an appropriate method of contraception during the observation period and for 8 weeks after the last dose of study drug.

13. Patients with HBV or HCV infection are required to be on antiviral therapy for the duration of the trial.

Subjects voluntarily enrolled in this study, signed informed consent, good compliance and cooperation with follow-up.

Exclusion Criteria:

- Patients will not be entered into this study if they meet any of the following criteria.

1. History of other malignancies within the previous 5 years or concurrently, except for cured basal cell carcinoma of the skin and carcinoma in situ of the cervix and papillary thyroid cancer
2. History of ruptured esophagogastric fundic varices, hepatic encephalopathy, massive ascites, and abdominal infection
3. Patients with previous use of other anti-angiogenic drugs, immunotherapeutic drugs, radiotherapy or systemic chemotherapy
4. Prior use of immunosuppressive drugs, excluding nasal spray and inhaled corticosteroids or physiologic doses of systemic steroids (i.e., no more than 10 mg days of prednisolone or equivalent pharmacologic doses of other corticosteroids), within 14 days prior to the first administration of kareolizumab
5. Known hypersensitivity to apatinib, carrilizumab, oxaliplatin, or drug excipients; or severe allergic reactions to other monoclonal antibodies
6. Live attenuated vaccines administered within 4 weeks prior to the first dose or scheduled to be administered during the study.
7. Known uncontrolled or symptomatic active central nervous system (CNS) metastases as evidenced by the presence of clinical signs, cerebral edema, spinal cord compression, carcinomatous meningitis, soft meningeal disease, and or progressive growth. Patients with a history of CNS metastases or spinal cord compression who are clearly treated and clinically stable after discontinuation of anticonvulsants and steroids for 4 weeks prior to the first dose of the study may be enrolled in the study.
8. The presence of > grade 1 peripheral neuropathy
9. The presence of any active autoimmune disease or a history of autoimmune disease
10. Presence of the following within 6 months prior to study entry: myocardial infarction, severe unstable angina, NYHA class 2 or higher cardiac insufficiency, poorly controlled arrhythmias (including QTcF intervals >450 ms in men and >470 ms in women, QTcF intervals calculated using the Fridericia formula), symptomatic congestive heart failure, cerebrovascular accident ( including transient ischemic attack or symptomatic pulmonary embolism).
11. Hypertension that is not well controlled with antihypertensive medication (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg).
12. Abnormal coagulation (INR > 1.5 or APTT > 1.5 x ULN) with bleeding tendency or on thrombolytic or anticoagulant therapy
13. Known hereditary or acquired bleeding and thrombotic tendencies, e.g., hemophilia, coagulation disorders, thrombocytopenia, hypersplenism, etc.
14. Presence of significant coughing up of fresh blood, or hemoptysis of half a teaspoon (2.5 ml) or more per day within 2 months prior to study entry
15. The presence of clinically significant bleeding symptoms or a definite bleeding tendency within 3 months prior to study entry, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, fecal occult blood +++ or more at baseline, or vasculitis
16. Arteriovenous thrombotic events such as cerebrovascular accidents (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism that occurred within 6 months prior to study entry
17. Known presence of hereditary or acquired bleeding and thrombotic tendencies (e.g. hemophiliacs, coagulation disorders, thrombocytopenia, hypersplenism, etc.)
18. The need for long-term anticoagulation therapy with warfarin or heparin, or the need for long-term antiplatelet therapy (aspirin ≥ 300 mg days or clopidogrel ≥ 75 mg days)
19. Concurrent severe infection (e.g., requiring intravenous antibiotics, antifungal or antiviral drugs) within 4 weeks prior to the first dose, or fever of unknown origin >38.5°C prior to the first dose during the screening period
20. Participation in any other drug clinical study within 4 weeks prior to the first dose, or no more than 5 half-lives from the last study dose
21. A known history of psychotropic substance abuse or drug use
22. The presence of other serious physical or mental illnesses or abnormal laboratory tests that may increase the risk of participation in the study or interfere with the results of the study, and patients who, in the opinion of the investigator, are not suitable for participation in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-05-06 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Major Pathological Response(MPR) 10% | Up to two years
  Survival tumor ≤10% during surgery

SECONDARY OUTCOMES:
ORR | Up to two years
  The proportion of patients with tumor size reduction of a predefined amount and for a minimum time period
1-year tumor recurrence-free rate RFS | Up to one years
  Subjects underwent radical resection from the start until the date of the first documented tumor into recurrence or death from any cause, whichever occurred first
Disease free survival (DFS) | Up to two years
  Time to disease progression or postoperative recurrence in subjects starting from radical postoperative resection, during the treatment period, and during the follow-up period
Intraoperative and postoperative complications | Up to two years
  Including bleeding volume and prolonged hospital stay

IPD SHARING:
Plan to Share IPD: No